CLINICAL TRIAL: NCT06325033
Title: Prospective Clinical Validation of the Eleveld Pharmacokinetic and Pharmacodynamic Model of Propofol for Procedural Sedation in Adults.
Brief Title: Prospective Validation of the Eleveld Model of Propofol for Procedural Sedation in Adults.
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: 18546
Record Dates: First submitted 2024-02-08; First posted 2024-03-22 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Deep Sedation
Keywords: Procedural sedation; Propofol; Validation; Eleveld model

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients age ≥ 18 - <65 and BMI <30: Adult patients for procedural sedation in the University Medical Center Groningen (UMCG) between 01-01-2024 and 01-01-2025.
- Patients age ≥ 18 - <65 and BMI ≥ 30: Adult patients for procedural sedation in the UMCG between 01-01-2024 and 01-01-2025.
- Patients age ≥ 65 and over: Adult patients for procedural sedation in the UMCG between 01-01-2024 and 01-01-2025.

SUMMARY:
The goal of this prospective observational study is to identify effect site concentrations (CET) of propofol using the Eleveld model for different levels of procedural sedation.

The main question it aims to answer is to identify CET propofol using the Eleveld model for different levels of procedural sedation as measured by the modified observer's assessment of alertness and sedation score (MOAAS) and EEG monitoring.

Participants vital signs will be monitored according to the departmental protocol. Sedation will be administered using Target-Controlled Infusion (TCI) of propofol (administered by effect-site TCI using the Eleveld model) and remifentanil (administered by effect site TCI using the Eleveld model). Target controlled infusion of propofol and remifentanil is according to the departmental protocol. The MOAAS score will be noted every 5 minutes or when the target effect site concentration of propofol is altered. Depth of sedation will also be monitored using a non-invasive BIS® monitor.

DETAILED DESCRIPTION:
Since 2012 procedural sedation practices in Dutch hospitals has taken a huge flight. Propofol is the preferred drug of choice for moderate to deep sedation. This can be titrated by using pharmacokinetic (PK) and pharmacodynamic (PD) models programmed in infusion pumps for target controlled infusion (TCI). Several pharmacokinetic-pharmacodynamic (PKPD) models for TCI propofol are available. While most TCI systems incorporate PK or PKPD models for specific patient groups such as adults, children or older patients, the Eleveld model has been developed for TCI of propofol for general anesthesia and sedation in a broad range of patients. In 2021 Vellinga et al published a study on the validation of the Eleveld model in patients undergoing general anesthesia. So far, the Eleveld model has not been externally validated for the use of procedural sedation in adult patients.

The aim of this study is to identify effect-site target concentrations of propofol for the Eleveld model that are associated with moderate to deep sedation levels, MOAAS 3-1 and the associated bispectral index ( BIS) levels in adult patients.

The secondary outcomes are: time to introduction of the endoscope and the time to reach MOAAS 5 after having stopped TCI propofol. The use of vasopressors such as ephedrine, phenylephrine or norepinephrine. The need for airway maneuvers such as chin lift, jaw thrust or nasopharyngeal airway.

The purpose of this investigation is to produce normalizing graphs of propofol drug infusion and TCI target concentrations for clinical sedation using the Eleveld TCI model. It mirrors the validation study of the Eleveld model. The sample size estimation of that study was determined by estimation bounds of the model-based drug concentration prediction accuracy. That study used 25 individuals for four groups: children, non-obese, elderly, and obese adults. Aside from the determination of prediction accuracy of the Eleveld model, an important secondary result was normalizing graphs of target concentrations, drug infusion, and drug effects in clinical practice.

The intention of the current investigation is to reproduce the normalizing graphs of TCI targets, drug infusion and effects similar to the Eleveld propofol TCI model validation study, but targeted to sedation rather than anesthesia. The current investigation uses no blood samples so sample size estimation cannot be based on model-based drug concentration prediction accuracy. We determined that a sample size similar to the validation study is appropriate and propose allocating 25 patients per group and three groups: non-obese, elderly and obese adults, for a total of 75 individuals.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients for procedural sedation in the UMCG between 01-01-2024 and 01-01-2025.

Exclusion Criteria:

* Age <18 years; use of esketamine during the procedure, use of benzodiazepines prior or during the procedure, hearing disability, BIS quality index < 50

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Three groups of 25 adult patients each, undergoing a diagnostic of interventional procedure at the endoscopy suite under procedural sedation.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2024-01-17 (Actual); Primary Completion 2024-07-11 (Actual); Study Completion 2024-07-11 (Actual)

PRIMARY OUTCOMES:
To identify effect-site target concentrations of propofol for the Eleveld model that are associated with moderate to deep sedation levels, MOAAS 3-1 and the associated BIS levels in adult patients. | From start of propofol infusion until end of propofol infusion, assessed for a maximum of 8 hours
  The intention of the current investigation is to reproduce the normalizing graphs of TCI targets, drug infusion and effects similar to the Eleveld propofol TCI model validation study, but targeted to sedation rather than anesthesia.

SECONDARY OUTCOMES:
Induction time | From start of propofol infusion until introduction of endoscope, assessed for a maximum of 20 minutes.tart of the sedation.
  Time from start of propofol infusion to introduction of the endoscope.
Recovery time | The time from stopping propofol infusion until reaching sedation and recovery level MOAAS 5 assessed or a maximum of up to 1 hour.
  The time to reach MOAAS 5 after having stopped target controlled infusion of propofol.
Adverse events | From start of propofol infusion until discharge from the recovery room, assessed for a maximum of 10 hours.
  The use of vasopressors such as ephedrine, phenylephrine or norepinephrine. The need for airway maneuvers such as chin lift, jaw thrust or nasopharyngeal airway.

CONTACTS AND LOCATIONS:
Overall Officials: Mendy Driesens, MSc, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Eleveld DJ, Colin P, Absalom AR, Struys MMRF. Pharmacokinetic-pharmacodynamic model for propofol for broad application in anaesthesia and sedation. Br J Anaesth. 2018 May;120(5):942-959. doi: 10.1016/j.bja.2018.01.018. Epub 2018 Mar 12. PMID 29661412
- [Result] Vellinga R, Hannivoort LN, Introna M, Touw DJ, Absalom AR, Eleveld DJ, Struys MMRF. Prospective clinical validation of the Eleveld propofol pharmacokinetic-pharmacodynamic model in general anaesthesia. Br J Anaesth. 2021 Feb;126(2):386-394. doi: 10.1016/j.bja.2020.10.027. Epub 2020 Dec 13. PMID 33317804
- [Result] Xi C, Sun S, Pan C, Ji F, Cui X, Li T. Different effects of propofol and dexmedetomidine sedation on electroencephalogram patterns: Wakefulness, moderate sedation, deep sedation and recovery. PLoS One. 2018 Jun 19;13(6):e0199120. doi: 10.1371/journal.pone.0199120. eCollection 2018. PMID 29920532

DOCUMENTS (1):
  • Study Protocol (2023-11-23): https://cdn.clinicaltrials.gov/large-docs/33/NCT06325033/Prot_000.pdf